CLINICAL TRIAL: NCT04647773
Title: A Multicenter, Randomized, Double-Blind, Double-Dummy, Placebo- and Pregabalin Capsule-Controlled, 13-Week, Adaptive-design Phase 2/3 Study to Evaluate the Efficacy and Safety of HSK16149 Capsules in Chinese Patients With Diabetic Peripheral Neuropathic Pain
Brief Title: To Evaluate the Efficacy and Safety of HSK16149 Capsule in Chinese Patients With Diabetic Peripheral Neuropathic Pain
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Haisco Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HSK16149-201/301
Record Dates: First submitted 2020-11-16; First posted 2020-12-01 (Actual); Last update posted 2020-12-01 (Actual); Status verified 2020-11

CONDITIONS: Diabetic Peripheral Neuropathic Pain
MeSH Terms: interventions — BID protein, human; Pregabalin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- HSK16149 20mg BID (Experimental)
  Interventions: Drug: HSK16149 20mg BID
- HSK16149 40mg BID (Experimental)
  Interventions: Drug: HSK16149 40mg BID
- HSK16149 60mg BID (Experimental)
  Interventions: Drug: HSK16149 60mg BID
- HSK16149 80mg BID (Experimental)
  Interventions: Drug: HSK16149 80mg BID
- Pregabalin 150mg BID (Active Comparator)
  Interventions: Drug: Pregabalin 150mg BID
- Placebo BID (Placebo Comparator)
  Interventions: Drug: Placebo BID

INTERVENTIONS:
Drug: HSK16149 20mg BID — HSK16149 20mg, orally twice a day, treatment period; 13-weeks fixed dose.
  Arms: HSK16149 20mg BID
Drug: HSK16149 40mg BID — HSK16149 40mg, orally twice a day, treatment period; 13-weeks fixed dose.
  Arms: HSK16149 40mg BID
Drug: HSK16149 60mg BID — HSK16149 60mg, orally twice a day, treatment period; 1-week titration and 12-weeks fixed dose.
  Arms: HSK16149 60mg BID
Drug: HSK16149 80mg BID — HSK16149 80mg, orally twice a day, treatment period; 1-week titration and 12-weeks fixed dose.
  Arms: HSK16149 80mg BID
Drug: Pregabalin 150mg BID — Pregabalin 150mg, orally twice a day, treatment period; 1-week titration and 12-weeks fixed dose.
  Arms: Pregabalin 150mg BID
Drug: Placebo BID — Placebo, orally twice a day, treatment period; 13-weeks fixed dose.
  Arms: Placebo BID

SUMMARY:
Investigate the efficacy and safety of HSK16149 capsules in Chinese diabetic peripheral neuropathic pain (DPNP) following 13 weeks treatment in comparison to placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent;
2. Males or females aged 18-75 years of age inclusive;
3. Diagnosis of diabetic peripheral neuropathic pain (DPNP) and diabetic peripheral neuropathy (DPN) pain ≥ 6 months;
4. HbA1c ≤ 9.0% at screening and on a stable antidiabetic medication regimen for at least 30 days prior to screening;
5. At Screening, pain scale (VAS) of ≥40 mm and <90 mm.

Exclusion Criteria:

1. Peripheral neuropathy or pain unrelated to DPN that may confuse the assessment of DPNP.
2. Skin conditions in the area affected by neurupathy that could alter sensation.
3. Chronic systemic diseases that may affect subjects' participation in the study.
4. Severe hematologic, hepatic or renal dysfunction, the subject will be excluded if:

   1. Neutrophils < 1.5 × 10^9/L, or platelet < 90 × 10^9/L, or hemoglobin < 100 g/L, or
   2. AST/ALT > 2.5 × upper limit of normal (ULN), or TBIL > 1.5 × ULN, or
   3. Estimation of glomerular filtration rate (eGFR) < 60 mL/min / 1.73 m^2, or
   4. Creatine kinase > 2.0 × ULN.
5. History of substance abuse or alcohol abuse.
6. Acute complications of diabetes in the 6 months prior to screening.
7. Any active infections at screening.
8. HBsAg or HCV Ab positive, or HIV Ab positive, or serum TP Ab positive.
9. Inability or unwillingness to discontinue any other prohibited concomitant medications (see Section 6.3).
10. Failure to response to previous treatment with pregabalin at doses ≥ 300 mg/d or gabapentin at doses ≥ 1200 mg/d for treatment of DPNP.
11. History of allergic or medically significant adverse reaction to investigational products or their excipients, acetaminophen or related compounds.
12. History of suicidal behavior or attempted suicide.
13. Pregnant or preparing for pregnancy or breastfeeding during the study period, or subjects were not willing to use reliable contraceptives methods from the date of ICF signature until 28 days after the last trial drug administration, or planning to use progesterone contraceptives during this period.
14. Participated in another clinical study within 30 days prior to screening.
15. Other conditions of the subjects who are unlikely to comply with the protocol.
16. Could potentially affect a subject's safety.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 687 (Estimated)
Dates: Start 2020-12-02 (Estimated); Primary Completion 2022-11-09 (Estimated); Study Completion 2022-11-16 (Estimated)

PRIMARY OUTCOMES:
Compare the change from baseline in Average Daily Pain Score（ADPS） between HSK16149 and placebo at week 5. | Baseline and week 5
  The mean change in average daily pain score (ADPS) was measured using a 11-point numeric rating scale (NRS; 0 [no pain] to 10 [worst possible pain]. The rating averaged over a 7-day period and was based on entries in patients' daily pain diaries.
Compare the change from baseline in Average Daily Pain Score （ADPS） between HSK16149 and placebo at week 13. | Baseline and week 13
  The mean change in average daily pain score (ADPS) was measured using a 11-point numeric rating scale (NRS; 0 [no pain] to 10 [worst possible pain]. The rating averaged over a 7-day period and was based on entries in patients' daily pain diaries.

SECONDARY OUTCOMES:
Compare the response rate between HSK16149 and placebo at week 5 (Proportion of subjects whose ADPS decreased by ≥30% and ≥50% from baseline ). | Baseline and week 5
  Ratio of Participants Responding to Treatment, as Measured by Average Daily Pain Score (ADPS) Reduction from Baseline. The ADPS is used to determine categorical response rates.
AE, laboratory tests, physical and neurological examination, vital signs and 12-lead ECG to evaluate the safety of HSK16149 in 5 weeks post treatment. | From week 1 to week 5
  Number and severity of AEs, clinical laboratory abnormalities, physical examinations, 12-lead electrocardiograms (ECGs), and vital signs.
Compare the response rate between HSK16149 and placebo at week 13 (Proportion of subjects whose ADPS decreased by ≥30% and ≥50% from baseline ). | Baseline and week 13
  Ratio of Participants Responding to Treatment, as Measured by Average Daily Pain Score (ADPS) Reduction from Baseline. The ADPS is used to determine categorical response rates.
Compare the change from baseline in ADPS between HSK16149 and placebo at week 1 to 13. | From week 1 to week 13
  The mean change in average daily pain score (ADPS) was measured using a 11-point numeric rating scale (NRS; 0 [no pain] to 10 [worst possible pain]. The rating averaged over a 7-day period and was based on entries in patients' daily pain diaries.
Compare the change from baseline in Visual Analog Scale （VAS） between HSK16149 and placebo at week 13. | Baseline and week 13
  VAS, in which the participant rates pain on a 100 mm-long horizontal line, where 0 mm = no pain and 100 mm = worst possible pain.
Compare the change from baseline in Short-Form McGill Pain Questionnaire (SF-MPQ) between HSK16149 and placebo at week 13. | Baseline and week 13
  Participants rate their pain in three parts of the questionnaire, which are combined into a single pain intensity score:
  Part 1 - fifteen descriptors of pain intensity, on a scale of 0 (none) to 3 (severe)
  Part 2 - a visual analog scale (VAS), in which the participant rates pain on a 100 mm-long horizontal line, where 0 mm = no pain and 100 mm = worst possible pain
  Part 3 - a Present Pain Intensity index in which the participant rates present pain intensity on a scale of 0 (no pain) to 5 (most intense pain)
Compare the Patient Global Impression of Change（PGIC） between HSK16149 and placebo at week 13. | Week 13
  Patient global impression of change (PGIC) on a 7-point categorical scale, where 1 = very much improved and 7 = very much worse.
Compare the change from baseline in Average Daily Sleep Interference score (ADSIS) between HSK16149 and placebo at week 13. | Baseline and week 13
  The sleep interference scores on a scale of 0-10, where 0 = pain did not interfere with sleep to 10 = pain completely interfered with sleep. The weekly ADSIS is based on participants daily sleep interference scores.
Compare the change from baseline in EuroQol-5-Domain-5-Level health questionnaire (EQ-5D-5L) between HSK16149 and placebo at week 13. | Baseline and week 13
  The change from baseline in total EuroQol-5-Domain-5-Level health questionnaire.
AE, laboratory tests, physical and neurological examination, vital signs and 12-lead ECG to evaluate the safety of HSK16149 during the trial. | From week 1 to week 14
  Number and severity of AEs, clinical laboratory abnormalities, physical examinations, 12-lead electrocardiograms (ECGs), and vital signs.
Pharmacokinetic (PK) characteristics of HSK16149 capsules in Chinese patients with diabetic peripheral neuropathic pain. | Week 1,week 5,week 11,week 13
  Pharmacokinetics will be determined by measuring serum concentration of HSK16149.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University First Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pan T, Ma J, Li Y, Wang K, Jiang C, Zhang Y, Liu J, Du R, Zhang W, Bian F, Zhang F, Wang L, Pang S, Ning T, Wang B, Li Y, Wu X, Zhang K, Tang X, Hu H, Sun X, Li P, Cheng Z, Sun J, Yang J, Wang Y, Gao J, Mao H, Li F, Huang Q, Li Y, Peng Z, Guo X. Rapid Onset of Pain Relief with Crisugabalin in Patients with Diabetic Peripheral Neuropathic Pain: Findings from a Multicenter, Randomized, Double-Blind, Controlled Study. Pain Ther. 2025 Aug;14(4):1311-1329. doi: 10.1007/s40122-025-00745-3. Epub 2025 May 16. PMID 40377855
- [Derived] Guo X, Zhang T, Yuan G, Zeng W, Hu Q, Ma J, Li Y, Li H, Zhang Y, Liu J, Bian F, Zhang W, Zhang F, Pang S, Li Y, Wu X, Tang X, Zhang K, Pan T, Hu H, Cheng Z, Wang Y, Gao J, Sun J. GABA Analogue HSK16149 in Chinese Patients With Diabetic Peripheral Neuropathic Pain: A Phase 3 Randomized Clinical Trial. JAMA Netw Open. 2024 Aug 1;7(8):e2425614. doi: 10.1001/jamanetworkopen.2024.25614. PMID 39158916